CLINICAL TRIAL: NCT01637025
Title: A Prospective, Randomized, Controlled Study to Evaluate the Safety and Effectiveness of Traumastem as an Adjunct to Hemostasis for Tissue Bleeding in Open Cardiac, Intra-abdominal (Including Retroperitoneal) and Pelvic Surgery
Brief Title: Oxidized Cellulose hEmostAsis evaluatioN
Acronym: OCEAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Baxter Innovations GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 621101
Record Dates: First submitted 2012-07-06; First posted 2012-07-10 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Intra-operative Bleeding

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Traumastem - oxidized cellulose strip (Experimental)
  Interventions: Device: Oxidized cellulose strip
- Surgicel® Original - oxidized regenerated cellulose strip (Active Comparator)
  Interventions: Device: Oxidized regenerated cellulose strip

INTERVENTIONS:
Device: Oxidized cellulose strip — Single use, intra-operative application to the target bleeding site
  Arms: Traumastem - oxidized cellulose strip
Device: Oxidized regenerated cellulose strip — A substance used to promote hemostasis (stops bleeding) based on oxidized regenerated cellulose
  Other Names: Tabotamp®
  Arms: Surgicel® Original - oxidized regenerated cellulose strip

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of Traumastem to help stop bleeding in participants undergoing open cardiac, intra-abdominal (including retroperitoneal) and pelvic surgery as compared to Surgicel® Original (Surgicel; in some countries marketed as Tabotamp®)

ELIGIBILITY:
INCLUSION CRITERIA AT SCREENING:

1. Participants and/or legal representative has/have provided signed informed consent. An assent form should be signed by Participants less than 18 years of age, if possible;
2. Participants undergoing planned (non-emergency) open cardiac, intra-abdominal (including retroperitoneal) and pelvic surgery;
3. Participants of childbearing potential present with a negative serum pregnancy test, and agree to employ adequate birth control measures for the duration of the study. Acceptable contraception methods are restricted to abstinence, barrier contraceptives, intrauterine contraceptive devices or licensed hormonal products;
4. Participants are willing and able to comply with the requirements of the clinical investigation plan (CIP).

   INCLUSION CRITERIA INTRA-OPERATIVE:
5. Soft tissue, vascular/anastomotic or parenchymal bleeding is present after primary surgical hemostasis has been achieved. The TBS is defined as intra-operative bleeding where conventional methods for achieving hemostasis are ineffective (based on the type of tissue) or impractical (based on the location) and where treatment with topical hemostatic adjuncts such as Traumastem is deemed appropriate for use.

EXCLUSION CRITERIA:

1. Emergency surgery;
2. Transplantation surgery;
3. Minimally invasive surgery;
4. Neurological and ophthalmological surgery;
5. Major arterial bleeding at the target bleeding site (TBS);
6. Major intra-operative complications that require resuscitation or deviation from the planned surgical procedure;
7. Severe local inflammation at the operating field;
8. Any prior radiation therapy to the operating field;
9. Known severe congenital or acquired immunodeficiency (eg, human immunodeficiency virus [HIV] infection or long-term [> 3 months] treatment with immunosuppressive drugs);
10. Known hypersensitivity to components of the investigational device;
11. Participant is pregnant or lactating at the time of enrollment or becomes pregnant prior to the planned surgery. If the participant becomes pregnant during the 30 days following treatment exposure, attempts will be made to follow her through completion of the pregnancy. The investigator will record a narrative description of the course of the pregnancy and its outcome;
12. Participant has a clinically significant medical, psychiatric, or cognitive illness, or drug/alcohol abuse that, in the opinion of the investigator, would affect participant's safety or compliance;
13. Participant has participated in another clinical study involving an investigational device/drug within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an investigational device/drug during the course of this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2012-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events (AEs)/ adverse device effects (ADEs) | ≤30 ± 5 days/ end-of-study visit after device application
  Occurrence of adverse events (AEs)/ adverse device effects (ADEs) up to 30 ± 5 days/ end-of-study visit after device application.

CONTACTS AND LOCATIONS:
Overall Officials: Edith Hantak, DVM, Study Director — Baxter Innovations GmbH
Locations (24):
- Czechia (7):
  - Chirurgicke oddeleni Nemocnice Liberec, Liberec
  - Kardiochirurgicke oddeleni FN Plzen, Plzen - Lochotin
  - Chirurgicka klinika FN KV, Prague
  - Chirurgicka klinika UVN, Prague
  - Chirurgicke oddeleni Fakultni nemocnice Na Bulovce, Prague
  - Kardiochirurgicka klinika FN KV, Prague
  - Klinika kardiovaskularni chirurgie IKEM, Prague
- Germany (6):
  - Klinik für Allgemein-, Visceral- und Transplantationschirurgie Charité Berlin, Berlin
  - Klinik für Allgemein-, Visceral-, Gefäß- und Thoraxchirurguie Charité Universitätsmedizin Berlin - Campus Mitte, Berlin
  - Allgemein- und Viszeralchirurgie Johann Wolfgang Goethe Universitätsklinikum, Frankfurt am Main
  - Klinik für Allgemeine Chirurgie, Viszeral-, Gefäß- und Kinderchirurgie Universitätsklinikum des Saarlandes, Homburg/Saar
  - Klinik für Allgemein- und Viszeralchirurgie Klinikum Magdeburg, Magdeburg
  - Klinik und Poliklinik für Allgemein- und Abdominalchirurgie Universitätsmedizin Mainz, Mainz
- Hungary (6):
  - I. Surgery Clinic Semmelweis Egyetem Általános Orvostudományi Kar, Budapest
  - Department of General Surgery Petz Aladár Megyei Oktató Kórház, Győr
  - Gynaecology and Obstetrics Petz Aldor Country Teaching Hospital, Győr
  - Department of General Surgery Békés Megyei Képviselotestület Pándy Kálmán Kórház, Gyula
  - Department of Surgery Albert Szentgyörgyi Clinical Center, Szeged
  - Department of General Surgery Békés Megyei Képviselotestület Pándy Kálmán Kórház, Székesfehérvár
- Poland (5):
  - Klinika Chirurgii Naczyniowej, Ogólnej i Angiologii, Samodzielny Publiczny Szpital Kliniczny Nr 2 PUM,, Szczecin
  - Klinika Chirurgii Ogólnej i Translantacyjnej, Samodzielny Publiczny Szpital Kliniczny Nr 2 PUM,, Szczecin
  - Niepubliczny Specjalistyczny Zakład Opieki Zdrowotnej "MEDICUS",, Środa Wielkopolska
  - Klinika Chirurgii Naczyniowej, Instytut Hematologii I Transfuzjologii,, Warsaw
  - Klinika Chirurgii Ogólnej, Gastroenterologicznej i Endokrynologicznej, Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wrocławiu, Wroclaw